CLINICAL TRIAL: NCT03405662
Title: Examining the Impact of Photobiomodulation on Cognition, Behavior, and Biomarkers of Alzheimer's Disease
Brief Title: Impact of Photobiomodulation (PBM) on Biomarkers of Alzheimer's Disease
Acronym: PBMbiomarker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OsherRAP
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants randomized to the "Active PBM" group will use an active Vielight Neuro device, for 16 weeks, once every other day (e.g., Mon, Wed, Fri) for 20 minutes.
  Participants randomized to the "Sham PBM" group will use a a sham Vielight Neuro device, for 16 weeks, once every other day (e.g., Mon, Wed, Fri) for 20 minutes.
  All study participants will undergo cognitive and behavioral assessments, blood draw, and lumbar puncture at baseline (before using Vielight Neuro Gamma device) and after 16 weeks of using the Vielight Neuro Gamma device.
  Upon completion of the post-16 week assessments, blood draw, and lumbar puncture, patients randomized to the Sham PBM group will be offered an opportunity to use an active Vielight Neuro Gamma device for 16 weeks. We will assess cognition and behavioral symptoms in Sham patients who opt to undergo active PBM 16 weeks after they start active PBM treatments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blind assignment determined by a computer-generated random allocation schedule
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acitve PBM (Active Comparator): This arm will receive active photobiomodulation (PBM), delivered with the Vielight Neuro Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes for 16 weeks.
  Interventions: Device: Vielight Neuro Gamma
- Sham PBM (Sham Comparator): This arm will not receive active photobiomodulation (PBM). Instead, they will use a sham Vielight Neuro Gamma device, once every other day (e.g., Mon, Wed, Fri) for 20 minutes for 16 weeks.
  Interventions: Other: Sham Vielight Neuro Gamma

INTERVENTIONS:
Device: Vielight Neuro Gamma — The Vielight Neuro Gamma is headset that delivers transcranial (through the scalp and skull) and intranasal (through the nose) near infrared (NIR) light. The device is engineered for increased efficacy and easy domestic use for comprehensive brain photobiomodulation (PBM). The NIR lights are pulsed at a 40 Hz rate, which correlates with electroencephalogram (EEG) gamma brain wave entrainment.
  Arms: Acitve PBM
Other: Sham Vielight Neuro Gamma — The Sham Vielight Neuro Gamma headset is identical to the active Vielight Neuro Gamma headset and intranasal light emitting diode (LED) except it has a power output of 0.
  Arms: Sham PBM

SUMMARY:
Photobiomodulation (PBM) describes the use of near-infrared light (which is not visible to the eye) to heal and protect tissue that has either been injured, is degenerating, or else is at risk of dying. Research suggests that the light delivered during PBM enhances the body's biochemical ability to store and use energy and increase blood flow, which triggers the body's natural healing processes. The primary goal of this study is to determine if PBM administered transcranially (through the scalp and skull) and intranasally (inside the nose) with a commercially available device is safe and tolerable for patients with mild-to-moderate Alzheimer's disease (AD). Secondary goals are to examine whether tPBM has an effect on cognitive function and behavioral symptoms in patients with AD and whether tPBM has an effect on fluid biomarkers of AD. A biomarker is a specific physical trait used to measure the progress of a disease or condition.

DETAILED DESCRIPTION:
Alzheimer's disease (AD), the most common form of dementia, is characterized by the loss of higher brain function such as memory, problem-solving abilities, and language. Photobiomodulation (PBM) describes a kind of light therapy that uses red or near-infrared light to stimulate, heal, regenerate, and protect tissue that has either been injured, is degenerating, or else is at risk of dying. The pathological hallmarks of AD include senile plaques rich in β-amyloid (Aβ) peptide and neurofibrillary tangles composed of hyperphosphorylated tau (p-tau). In animal models of AD, PBM reduces the size and number of brain Aβ plaques, p-tau, and neurofibrillary tangles. PBM also mitigates behavioral deficits in transgenic AD mouse models and humans with dementia. The goal of this sham-controlled pilot trial is to investigate the effects of PBM on the cognitive function, behavioral symptoms, and fluid (i.e., cerebrospinal fluid (CSF) and blood) biomarkers of AD pathology including amyloid burden, tangle pathology, axonal injury, microglia activation/inflammation, and neurotrophic factors in 16 patients with biomarkers-supported probable Alzheimer's dementia, according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.

The main goal of the study is to examine the safety and tolerability of home administered transcranial photobiomodulation (tPBM) with a commercially available device in patients with mild-to-moderate AD. Another goal of the study is to examine the effect PMB on cognitive function and behavioral symptoms in patients with probable AD. The study's final goal is to examine the effects of 16 weeks of PBM on fluid biomarkers of inflammation (i.e., monocyte chemoattractant protein 1 and 3 [MCP-1 and MCP-3] and macrophage inflammatory protein 1β [MIP-1β]), neurodegeneration (i.e., ubiquitin carboxyl-terminal hydrolase isozyme L1 [UCH-L1] and neurofilament light chain [NfL]) and neurotrophic factors (i.e., vascular endothelial growth factor [VEGF] and brain-derived neurotrophic factor [BDNF]). We will also explore the relationship between cognitive and behavioral changes after 16 weeks of PBM with changes in biomarkers of inflammation, neurotrophic factors, and neurodegeneration.

Sixteen patients with biomarkers-supported probable Alzheimer's dementia will be enrolled and randomly assigned to an active or sham PBM group. All patients will be asked to use the Vielight Neuro Gamma (real or sham) device for 20 minutes/day, every other day, for 16 weeks. Randomization with blind assignment will be determined by a computer-generated random allocation. We will assess safety and tolerability by comparing adverse events (AD) in each group. Cognition, behavioral symptoms, and biomarker measures will be assessed in all study participants at baseline and after 16 weeks of PBM. Biomarkers will be obtained through a blood draw and lumbar puncture. A lumbar puncture (also called a spinal tap) is a procedure to collect cerebrospinal fluid, or CSF), which surrounds the brain and spinal cord. During a lumbar puncture, a needle is carefully inserted into the spinal canal low in the back (lumbar area).

Study partners (e.g., caregivers) will be asked to answer questions about the study participant's memory and daily functioning at baseline and after 16 weeks of PBM. Study partners will also be trained and ask to help the study partners administer PBM treatments with the Vielight Neuro Gamma device at home for 16 weeks.

ELIGIBILITY:
Inclusion Criteria (for participants with AD):

* Diagnosis of AD supported by AD biomarkers (CSF or amyloid PET)
* Mini-Mental State Exam (MMSE) score > 13
* fluent in English
* has a reliable caregiver/study partner who can help administer and log PBM use
* no history of stroke or seizures
* willing to undergo 2 lumbar punctures approximately 4 months apart
* legally authorized representative consent

Exclusion Criteria: (for participants with AD)

* lack of assent to study procedures
* terminal illness (i.e., life expectancy < 1 year)
* started dementia medication (i.e., cholinesterase inhibitor or memantine) within the past 3 months or planning to start new dementia medication
* current participation in another research study that could potentially confound current study (e.g., medication or behavioral intervention)
* MMSE < 13
* history of structural brain lesions or stroke temporally related to the onset or worsening of cognitive impairment
* history of head trauma associated with injury-onset cognitive complaints or loss of consciousness for 10 minutes or longer.

Inclusion Criteria (for study partners):

* ability to answer questions about the primary participant's memory, behaviors, and activities of daily living
* willingness to help primary participant use and log the use of the Vielight Neuro Gamma device every other day for 16 weeks
* fluent in English

Exclusion Criteria (for study partners):

* major neurological or psychiatric condition
* terminal illness (i.e., life expectancy < 1 year)
* evidence of cognitive impairment
* inability to consent to study procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Chao, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - VA Health Care System, San Francisco, California
  - UCSF Memory and Aging Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Taboada L, Yu J, El-Amouri S, Gattoni-Celli S, Richieri S, McCarthy T, Streeter J, Kindy MS. Transcranial laser therapy attenuates amyloid-beta peptide neuropathology in amyloid-beta protein precursor transgenic mice. J Alzheimers Dis. 2011;23(3):521-35. doi: 10.3233/JAD-2010-100894. PMID 21116053
- [Background] Purushothuman S, Johnstone DM, Nandasena C, Mitrofanis J, Stone J. Photobiomodulation with near infrared light mitigates Alzheimer's disease-related pathology in cerebral cortex - evidence from two transgenic mouse models. Alzheimers Res Ther. 2014 Jan 3;6(1):2. doi: 10.1186/alzrt232. eCollection 2014. PMID 24387311
- [Background] Berman MH, Halper JP, Nichols TW, Jarrett H, Lundy A, Huang JH. Photobiomodulation with Near Infrared Light Helmet in a Pilot, Placebo Controlled Clinical Trial in Dementia Patients Testing Memory and Cognition. J Neurol Neurosci. 2017;8(1):176. doi: 10.21767/2171-6625.1000176. Epub 2017 Feb 28. PMID 28593105
- [Background] Sommer AP, Bieschke J, Friedrich RP, Zhu D, Wanker EE, Fecht HJ, Mereles D, Hunstein W. 670 nm laser light and EGCG complementarily reduce amyloid-beta aggregates in human neuroblastoma cells: basis for treatment of Alzheimer's disease? Photomed Laser Surg. 2012 Jan;30(1):54-60. doi: 10.1089/pho.2011.3073. Epub 2011 Oct 26. PMID 22029866
- [Background] Grillo SL, Duggett NA, Ennaceur A, Chazot PL. Non-invasive infra-red therapy (1072 nm) reduces beta-amyloid protein levels in the brain of an Alzheimer's disease mouse model, TASTPM. J Photochem Photobiol B. 2013 Jun 5;123:13-22. doi: 10.1016/j.jphotobiol.2013.02.015. Epub 2013 Mar 22. PMID 23603448

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-three (23) participants signed informed consent forms/were enrolled in the study. Nine (9) of these participants did not meet study inclusion criteria (e.g., baseline MMSEs were too low, or did not have AD biomarkers). Fourteen (14) participants were randomized: 7 to Active PBM; 7 to Sham PBM.
Period: Overall Study
Arm/Group | Acitve PBM | Sham PBM
Started | 7 | 7
Completed | 6 | 4
Not Completed | 1 | 3
Not completed — COVID-19 restriction | 1 | 0
Not completed — unblinding | 0 | 1
Not completed — placement in memory care facility | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acitve PBM | Sham PBM | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Full Range); unit: years] | 68.1 [54 to 85] | 72.4 [61 to 80] | 70.3 [54 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Mini-Mental State Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The MMSE ranges from 0 to 30. Higher scores are better.
  units on a scale | 23.4 (7.1) | 21.6 (4.4) | 22.5 (5.7)
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) [Mean (Standard Deviation); unit: units on a scale] — The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia. It is one of the most widely used cognitive scales in clinical trials and is considered to be the "gold standard" for assessing antidementia treatments. Scores (errors) on single scale range from 0 to 70. Higher scores are indicative of greater cognitive impairment.
  units on a scale | 35.5 (8.3) | 27.5 (20.0) | 31.5 (15.3)
Neuropsychiatric Inventory (NPI) [Mean (Standard Deviation); unit: units on a scale] — The Neuropsychiatric Inventory (NPI) measures the presence and severity of 12 neuropsychiatric symptoms. Symptoms are rated in terms of frequency (1=rarely, <1x/week; 2=sometimes, ~1x/week; 3=often, several times/week; and 4=very often, >1x/day) and severity (1=mild; 2=moderate; 3=severe). The composite symptom domain score (frequencyXseverity) ranges from 0 (no behavioral symptoms) to 144 points. Caregiver distress is rated for each positive neuropsychiatric symptom domain (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=very severe distress).
  units on a scale | 42.0 (29.8) | 21 (50.7) | 31.5 (41.5)
Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-ADL) [Mean (Standard Deviation); unit: units on a scale] — The ADCS-ADL assesses the competence of patients with dementia in basic and instrumental activities of daily living (ADLs). It can be completed by a caregiver in questionnaire format, or administered by a clinician/researcher as a structured interview. The ADCS-ADL is a 23 item scale that includes 6 basic activities of daily living items (e.g., grooming/dressing) and 17 instrumental activities of daily living items (e.g., cooking/managing finance) that provide a total score from 0-78, with a lower score indicating greater severity.
  units on a scale | 57.0 (7.5) | 68.4 (8.2) | 62.7 (9.6)
Color Trails Test (CTT), 1 [Mean (Standard Deviation); unit: seconds] — The Color Trails Test (CTT) is a neuropsychological test that assesses frontal and executive functioning, while minimizing the cultural and language barriers inherent in similar measures such as the traditional Trail Making Test. For test 1, the participant uses a pencil to rapidly connect circles numbered 1 through 25 in sequence.
  seconds | 114.1 (64.7) | 69.4 (33.0) | 95.5 (56.7)
CTT2 [Mean (Standard Deviation); unit: seconds] — The Color Trails Test (CTT) is a neuropsychological test that assesses frontal and executive functioning, while minimizing the cultural and language barriers inherent in similar measures such as the traditional Trail Making Test. For test 2, the participant rapidly connects numbered circles in sequence, alternating between two different colors.
  seconds | 248.3 (57.6) | 147.8 (75.4) | 206.4 (80.9)
CTT2/CTT1, index [Mean (Standard Deviation); unit: ratio] — The index is a ratio of the time it takes to complete the Color Trails Test (CTT) 2 over the time it takes to complete the CTT 1. The index provides a method for partialling out the effects of undivided attention and simple perceptual tracking on the alternating demands of CTT-2. Higher index scores indicate greater interference, less cognitive flexibility.
  ratio | 2.0 (1.2) | 1.2 (0.9) | 1.6 (1.1)
Plasma Aβ40 [Mean (Standard Deviation); unit: pg/mL] — Aβ40 is a 40 amino acid proteolytic product from the amyloid precursor protein (APP) that has gained attention as a biomarker correlating with Alzheimer disease (AD) onset, mild cognitive impairment, vascular dementia, and other cognitive disorders.
  pg/mL | 223.2 (74) | 219.0 (9) | 220.3 (55)
Plasma Aβ42 [Mean (Standard Deviation); unit: pg/mL] — Aβ42 is the 42 amino acid form of amyloid-β that plays a key role in the pathogenesis of Alzheimer's disease (AD) and is considered a core biomarker for the diagnosis of AD.
  pg/mL | 21.3 (6) | 20.0 (3) | 20.7 (5)
Plasma Aβ 42/40 [Mean (Standard Deviation); unit: ratio] — Decreased ratio of Aβ 42/40 is a strong marker of Alzheimer's disease and can be detected early in the disease progression, even before clinical dementia occurs.
  ratio | 0.08 (0.01) | 0.08 (0.01) | 0.08 (0.01)
Plasma tau [Mean (Standard Deviation); unit: pg/mL] — Tau is a microtubule-associated protein that forms insoluble filaments that accumulate as neurofibrillary tangles in Alzheimer's disease (AD).
  pg/mL | 1.6 (0.3) | 1.4 (0.3) | 1.5 (0.4)
Plasma P-tau181 [Mean (Standard Deviation); unit: pg/mL] — Tau phosphorylated at threonine 181 (p-tau181) is a highly specific biomarker for Alzheimer's disease pathology. Concentrations of P-tau181 might be increased in Alzheimer's disease (AD).
  pg/mL | 5.9 (1.5) | 5.2 (1.7) | 5.7 (1.6)
Plasma neurofilament light chain (NfL) [Mean (Standard Deviation); unit: pg/mL] — Neurofilament light chain (NfL) is a neuronal cytoplasmic protein highly expressed in large myelinated axons. Its levels increase in cerebrospinal fluid (CSF) and blood proportionally to the degree of axonal damage in a variety of neurological disorders, including Alzheimer's disease.
  pg/mL | 14.3 (5) | 17.2 (4) | 15.8 (5)
Plasma glial fibrillary acidic protein (GFAP) [Mean (Standard Deviation); unit: pg/mL] — Glial fibrillary acidic protein (GFAP) is a monomeric intermediate filament protein found in the astroglial cytoskeleton. This protein is not routinely secreted in blood or CSF and is only released after cell death or injury.
  pg/mL | 262.5 (79) | 276.4 (96) | 269.5 (88)
cerebrospinal fluid (CSF) Aβ40 [Mean (Standard Deviation); unit: pg/mL x 10^3] | 26.7 (9) | 20.4 (7) | 23.6 (8)
CSF Aβ42 [Mean (Standard Deviation); unit: pg/mL x 10^3] | 3.4 (2) | 1.9 (0.6) | 2.7 (1.4)
CSF Aβ42/40 [Mean (Standard Deviation); unit: ratio] | 0.1 (0.1) | 0.1 (0.02) | 0.1 (0.07)
CSF tau [Mean (Standard Deviation); unit: pg/mL] | 505 (323) | 382 (322) | 444 (319)
CSF P-tau181 [Mean (Standard Deviation); unit: pg/mL] | 439 (194) | 335 (202) | 388 (199)
CSF neurofilament light chain (NfL) [Mean (Standard Deviation); unit: pg/mL x 10^3] | 3.4 (1) | 3.3 (2) | 3.4 (2)
CSF glial fibrillary acidic protein (GFAP) [Mean (Standard Deviation); unit: pg/mL x 10^3] | 50.1 (43) | 54.2 (36) | 52.2 (40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog)
Description: The ADAS-cog is the most popular cognitive testing instrument used in clinical trials of nootropics. It consists of 11 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD. Higher ADAS-cog scores indicate greater cognitive impairment.
  The changes score was determined by calculating the ratio of the ADAS-cog score at week 16 over the ADAS-cog score at baseline. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in ADAS-cog score compared to baseline.
Time Frame: Baseline to 16 weeks
Population: One Active PBM patient did not return for post-treatment assessment due to pandemic-related lock-down. Two Sham PBM patients did not return for post-treatment assessment due to worsening of symptoms that necessitated placement in memory care facility. One Sham PBM patient was excluded due to unblinding.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 6 | 4
Ratio | 0.94 (0.2) | 1.4 (0.2)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.07, non-parametric Kolmogorov-Smirnov test

2. Secondary Outcome: Change in Performance on Color Trails Test (CTT2/CTT1 Index)
Description: CTT is a non-verbal test of visual attention, graphomotor sequencing, and effortful executive processing abilities (i.e., sustained attention and set shifting). A higher index score indicates less cognitive flexibility, a lower ability to shift attention.
Time Frame: Baseline to 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 6 | 4
Ratio | 1.1 (1) | 1.2 (0.08)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.29, non-parametric Kolmogorov-Smirnov test

3. Secondary Outcome: Change on the Neuropsychiatriac Inventory (NPI)
Description: NPI is a well-validated, reliable, multi-item instrument to assess psychopathology (e.g., behavioral symptoms) in AD based on a questionnaire completed by the participants' study partners. Higher scores indicate more symptoms and/or more severe symptoms.
  The changes score was determined by calculating the ratio of the week 16 NPI score over the baseline NPI score. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in NPI compared to baseline.
Time Frame: Baseline to 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 6 | 4
Ratio | 1.1 (2.2) | 1.87 (0.5)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.07, non-parametric Kolmogorov-Smirnov test

4. Secondary Outcome: Change on the Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL)
Description: ADCS-ADL assesses the competence of patients with AD in basic and instrumental activities of daily living (ADLs). It can be completed by a caregiver in questionnaire format, or administered by a clinician/researcher as a structured interview with a caregiver. ADCS-ADL scores range from 0-53, with higher scores indicating greater independence. The changes score was determined by calculating the ratio of the week 16 ADCS-ADL score over the baseline ADCS-ADL score. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in ADCS-ADL compared to baseline.
Time Frame: Baseline to 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 6 | 4
Ratio | 1.0 (2.2) | 0.9 (0.07)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.23, non-parametric Kolmogorov-Smirnov test

5. Secondary Outcome: Change in Plasma Levels of Aβ42
Description: Although Aβ42 is present in plasma, it is unclear whether it originates from peripheral sources or from the brain. Because Aβ can be transported bidirectionally across the blood-brain barrier, it has been hypothesized that there may be an equilibrium between CSF and plasma pools of Aβ. Decreased levels of Aβ42 in CSF occurs in conjunction with cognitive decline. However, patients with mutations in chromosome 21 that cause early-onset familial AD and patients with trisomy 21 have increased levels of plasma Aβ42 before the onset of the symptoms of dementia. Therefore, it is possible that plasma Aβ42 levels increase with cognitive decline. The change score was determined by calculating the ratio of plasma Aβ42 at week 16 over the ADAS-cog score at baseline.
Time Frame: Baseline to 16 weeks
Population: One Active REAL PBM patient did not return for post-treatment assessment due to pandemic-related lock-down; another REAL PBM patient's post-treatment sample was contaminated. One SHAM patient was excluded for unblinding, two SHAM patients were institutionalized during the study; two other SHAM patients had failed lumbar punctures.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 5 | 2
Ratio | 0.92 (0.1) | 1.0 (0.1)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.68, non-parametric Kolmogorov-Smirnov test

6. Secondary Outcome: Change in CSF Levels of Aβ42.
Description: Aβ42 is a biomarker of AD pathology. CSF levels of Aβ42 decrease in conjunction with the cognitive decline. The change score was determined by calculating the ratio of CSF Aβ42 at week 16 over the ADAS-cog score at baseline. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in CSF levels of Aβ42 compared to baseline.
Time Frame: Baseline to 16 weeks
Population: One Active REAL PBM patient did not return for post-treatment assessment due to pandemic-related lock-down; two REAL PBM patient's post-treatment samples were contaminated. One SHAM patient was excluded for unblinding, two SHAM patients were institutionalized during the study; two other SHAM patients had failed lumbar punctures.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 4 | 2
Ratio | 0.4 (0.1) | 1.3 (0.3)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.13, non-parametric Kolmogorov-Smirnov test

7. Secondary Outcome: Change in Plasma Levels of Tau.
Description: Tau, the microtubule-associated protein, forms insoluble filaments that accumulate as neurofibrillary tangles in Alzheimer's disease (AD). Research suggests that plasma tau levels increased with AD severity. The change score was determined by calculating the ratio of the week 16 plasma tau over the baseline plasma tau levels. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in plasma tau compared to baseline.
Time Frame: Baseline to 16 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 5 | 2
Ratio | 0.7 (0.2) | 1.0 (0.1)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.32, non-parametric Kolmogorov-Smirnov test

8. Secondary Outcome: Change in CSF Levels of Tau
Description: Tau forms insoluble filaments that accumulate as neurofibrillary tangles in AD. Increased levels of tau in CSF is a key characteristic of AD and is considered to result from neurodegeneration. The change score was determined by calculating the ratio of week 16 CSF tau over baseline CSF tau. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in CSF tau compared to baseline.
Time Frame: Baseline to 16 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 4 | 2
Ratio | 0.7 (0.5) | 1.1 (0.3)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.68, non-parametric Kolmogorov-Smirnov test

9. Secondary Outcome: Change in Plasma Levels of Neurofilament Light Chain (NfL)
Description: Neurofilament light chain (NfL) is a marker of axonal degeneration and is robustly elevated in the blood of many neurological and neurodegenerative conditions, including AD. The change score was determined by calculating the ratio of week 16 plasma levels of NfL over the baseline levels of plasma NfL. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in plasma levels of NfL compared to baseline.
Time Frame: Baseline to 16 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 5 | 2
Ratio | 1.0 (0.2) | 1.2 (0.4)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.86, non-parametric Kolmogorov-Smirnov test

10. Secondary Outcome: Change in CSF Levels of NfL
Description: Neurofilament light chain (NfL) is a marker of axonal degeneration and is robustly elevated in the blood of many neurological and neurodegenerative conditions, including AD. There is a strong relationship with cerebrospinal fluid (CSF) NfL, suggesting that these biomarker modalities reflect the same pathological process. The change score was determined by calculating the ratio of week CSF NfL over baseline CSF NfL. Thus, a change score of 1 signifies no change compared to baseline and change scores < 1 or > 1 reflect a decrease or an increase in CSF NfL compared to baseline.
Time Frame: Baseline to 16 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Acitve PBM | Sham PBM
Number analyzed (Participants) | 4 | 2
Ratio | 0.6 (0.3) | 0.7 (0.06)
Statistical Analysis 1: Comparison: Acitve PBM vs Sham PBM; Test type: Superiority; p = 0.32, non-parametric Kolmogorov-Smirnov test

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Acitve PBM | Sham PBM
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acitve PBM (N=7) | Sham PBM (N=7)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Disorientation (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyponatremia (General disorders) | 1 (1) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 1 (1)
Syncope (General disorders) | 1 (1) | 1 (1)
temporary device malfunction (Product Issues) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03405662/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03405662/ICF_001.pdf